CLINICAL TRIAL: NCT04506515
Title: Psychological Impact of COVID-19 Pandemic in Healthcare Workers in Spain: A Cross-sectional Study. PSIMCOV Group
Brief Title: Psychological Impact of COVID-19 Pandemic in Healthcare Workers
Acronym: PSIMCOV
Status: Completed | Type: Observational
Sponsor: Hospital General Universitario de Valencia (Other)
Responsible Party: Principal Investigator, Carolina Soledad Romero Garcia, MD, PhD, Anesthesia and Critical care consultant, Hospital General Universitario de Valencia
Other Study IDs: COV2-2020
Record Dates: First submitted 2020-08-03; First posted 2020-08-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Covid19; Stress, Psychological; Work Related Stress; Epidemic Disease; SARS-CoV Infection
MeSH Terms: conditions — COVID-19; Stress, Psychological; Occupational Stress; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Psychological stress and adaptation at work score (PSAS) — completing a survey based on PSAS

SUMMARY:
Background. The current coronavirus disease (COVID-19) has a great impact worldwide. Healthcare workers play an essential role and are one of the most exposed groups.Information about the psychosocial impact on healthcare workers is limited.

Methods. 3109 healthcare workers completed a national, internet-based, cross-sectional 45-item survey between 9 and 19 April 2020. The objective is to assess the psychological impact of the COVID-19 pandemic in Spanish healthcare workers. A Psychological Stress and Adaptation at work Score (PSAS) was defined combining four modified versions of validated psychological assessment tests (A) Healthcare Stressful Test, (B) Coping Strategies Inventory,(C) Font-Roja Questionnaire and (D) Trait Meta-Mood Scale.

DETAILED DESCRIPTION:
PSAS (Psychological Stress and Adaptation at work Score) is a self conducted questionnaire designed to assess psychological impact in healthcare workers to match times of crisis and when the time is scarce. PSAS has a range between 0 and 105, and higher scores represent higher stress detected.

ELIGIBILITY:
Inclusion Criteria:

* Active healthcare workers in any private/public hospital > 18 years old

Exclusion Criteria:

* Refusal to participate

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Respondents are healthcare workers in any center/hospital treating patients and are involved directly or indirectily with patients who suffer from COVID-19.
  Respondents might be physicians, nurses, ancillary staff, etc or be involved in other type of jobs like administration, techinical support, kitchen and cleaning servicies, etc.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2020-04-19 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
PSAS (Psychological Stress and Adaptation at work Score) during the crisis | during the pandemic (April 9, 2020 to April 19, 2020)
  evaluate the severity of psychological impact of the pandemic in Spain in healthcare workers

SECONDARY OUTCOMES:
PSAS (Psychological Stress and Adaptation at work Score) in basal conditions | After the pandemic (back to regular activity to be considered in the future as we do not know it yet. It expected to be in less than one year.
  evaluate the psychological stress in Spain in healthcare workers

CONTACTS AND LOCATIONS:
Locations (1):
- CHGUV, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The investigators did not ask to the ethical committee board for data sharing approval

REFERENCES:
- [Background] Romero CS, Delgado C, Catala J, Ferrer C, Errando C, Iftimi A, Benito A, de Andres J, Otero M; PSIMCOV group*. COVID-19 psychological impact in 3109 healthcare workers in Spain: The PSIMCOV group. Psychol Med. 2022 Jan;52(1):188-194. doi: 10.1017/S0033291720001671. Epub 2020 May 14. PMID 32404217